CLINICAL TRIAL: NCT01641679
Title: Recurrent Differentiated Thyroid Cancer: Towards Personalized Treatment Based on Evaluation of Tumor Characteristics With PET (THYROPET
Brief Title: PET Evaluation of Recurrent Differentiated Thyroid Cancer
Acronym: THYROPET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: NL37266.031.11; M11TRP (Other: PTC NKI-AVL)
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Thyroid Neoplasms; Differentiated Thyroid Cancer
Keywords: Recurrent differentiated thyroid cancer; I124-PET/CT; FDG-PET/CT
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected recurrent DTC: 100 patients with biochemically suspected recurrent DTC

SUMMARY:
After initial treatment of differentiated thyroid cancer patients (DTC) are followed by a blood test, a biomarker called thyroglobulin, in order to detect a possible recurrence. Nowadays patients are treated 'blindly' with high dose radioactive iodine to treat a suspected recurrence. However, the scan made after therapy to verify the effect of the treatment shows that in up to 50% the treatment could be considered as futile.

124I - a radioactive isotope - in combination with whole body PET became recently available for use in the follow-up of DTC. This could make it possible before the therapy with high dose radioactive iodine to determine the extensiveness of the disease and whether effect of the therapy could be expected. Additionally, recurrent DTC lesions that do not accumulate iodine can be found without the futile treatment with 131I. FDG-PET (another PET modality) is able to detect these lesions. The value of FDG-PET before 131I treatment however has not been tested.

The combination of these two diagnostic tools, 124I-PET and FDG-PET, has a potential to allow earlier and better restaging and selection for treatment

DETAILED DESCRIPTION:
Differentiated thyroid cancer (DTC) is the most frequent endocrine tumor, with an annual incidence per 100.000 individuals of 1 - 3 in men and 2 - 4 in women. In general DTC has a good prognosis, and only 6% of patients will die of their disease, but the prognosis is less favourable when the disease recurs after primary treatment.

Measurement of the tumor marker Thyroglobulin (Tg) in serum plays a pivotal role in the follow-up of differentiated thyroid cancer. Serum Tg should be undetectable in DTC patients following thyroid remnant ablation with radioactive iodine-131 (131I), and any detectable level signals the persistence of (neoplastic) thyroid tissue. A serum Tg cut-off level of ≥ 2 ng/ml following rhTSH is highly sensitive for identifying patients in whom persistent tumor may be found.

Historically the follow-up of patients with DTC included diagnostic planar scintigraphy with a low dose of 131I, but nowadays this is no longer recommended because of poor sensitivity. Instead, whole body scintigraphy after blind administration of high dose, 'therapeutic', 131I is recommended, both to diagnose and stage the potential recurrence, and to initiate its treatment. This strategy can be effective, but an estimated 38% - 50% of patients will have a negative post-therapeutic whole body scan and/or no objective therapy effect. These patients will have received a total body irradiation of 450 mSv and potentially will have suffered from side effects such as nausea, sialoadenitis, loss of taste, or reduced spermatogenesis. Also, the prolonged thyroid hormone withdrawal and subsequent hypothyroidism necessary for 131I therapy has major impact on quality of life with a majority of patients suffering from significant changes in physical, psychological, and social well-being. The high frequency of high dose 131I therapies from which patients do not derive any benefit but are exposed to its toxicity and potential adverse oncological effects, has led to a search for new diagnostic tools to improve the selection of patients before such treatment.

Historically, ultrasound of the neck is applied to detect local recurrence or regional lymph node metastases, and it allows direct biopsy to confirm the diagnosis. But ultrasound is limited to the neck only, and when it is negative in the presence of detectable Tg, a form of whole body evaluation is required.

Recently Iodine-124 (124I) became available as a novel radionuclide for whole body PET imaging in the follow-up of DTC, with a promising diagnostic accuracy and a considerably lower radiation exposure as compared to planar whole body scintigraphy after high dose 131I. Furthermore, recent experience has shown that 124I-PET images may be representative for the biodistribution and radiation dosimetry of subsequent treatment with high dose 131I. Thus, with the availability of 124I-PET, it might become possible to more accurately re-stage patients in a whole body procedure, perform dosimetry for subsequent 131I therapy and predict the outcome of the treatment.

At the same time, some recurrent DTC lesions do not accumulate iodine, which is correlated with tumor dedifferentiation and poor prognosis. Patients suspected of non-iodine accumulating DTC, so far only evident after futile blind 131I therapy, require restaging before local or systemic therapy may be installed. Metabolic PET imaging with the glucose analogon 18F-fluorodeoxyglucose (FDG), stimulated with rhTSH, has a high sensitivity for recurrent DTC in patients with detectable Tg and negative iodine scintigraphy, may correlate with a more aggressive tumor behaviour and poor prognosis, and is able to select patients for additional surgery or external beam radiotherapy. This technique is currently applied only when prior treatment and imaging with high dose 131I has proven to be ineffective. The value of FDG-PET before 131I treatment has not been tested.

The uptake of 124iodine and FDG are related to histopathological characteristics of tumor tissue, such as the resected primary tumor or metastases. 124I uptake is related to expression of the sodium iodine symporter (NIS), while FDG uptake is related to hexokinase-I (HKI) activity. The power of combined 124I-PET and FDG-PET for detection and characterization of DTC lesions has been suggested in proof of concept studies. The relation of these imaging findings and histopathological parameters (such as thyroglobulin, TTF1, Ki-67 and Cytokeratine-19 staining) and response to 131I treatment has not been elucidated in sufficiently large series.

Based on the characteristics of 124I-PET and FDG-PET, it is reasonable to assume that a combined strategy of imaging and histopathological evaluation at the time of suspected recurrence will yield adequate information on the disease stage prior to treatment with 131I, regardless of tumor dedifferentiation, with a potential impact on clinical decision making. This hypothesis needs proper testing, to increase fundamental knowledge about DTC and further improve treatment.

The multi-center design of this study requires a standard acquisition of the 124I-PET scans. Previously this was done for FDG-PET in the Netherlands, the so-called NEDPAS protocol. In order to compare the scans between the centers calibration and standardization of the 124I-PET scans prior to the start of the study will be done.

Additional to this objective the study aims to answer whether thyroid hormone withdrawal and rhTSH preparation for the 124I-PET results in different scan results.

In summary, high dose 131I treatment for recurrent DTC is effective in many cases, but the current blind approach also leads to overtreatment, delay, and unnecessary decrease in quality of life in a significant number of cases. As we have shown, a combination of diagnostic tests has a potential to allow earlier and better restaging and selection for treatment. The proposed trial aims to test the value and optimal implementation of these new tests, standalone and in combination, to derive parameters for a new personalised strategy for diagnosis and treatment of patients with (suspected) recurrent DTC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of differentiated thyroid cancer
* After complete thyroidectomy and ablation of functional remnants with 131I.
* Planned for blind high dose 131I treatment based on biochemically suspected recurrence, defined as a Tg-level above 2.0 ng/ml.
* Ultrasonography of the neck performed < 2 months prior to inclusion.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Incapacitated subjects
* Contrast enhanced CT performed < 4 months prior to inclusion
* I-131 therapy performed < 12 months prior to inclusion
* Indication for other therapy modality (ie. surgery in case of a positive ultrasonography, radiotherapy, embolization or chemotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with a history of DTC treated with total thyroidectomy and ablation who now have a suspicion of recurrence outside the neck based on a raised Tg and a negative neck ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The number of futile high-dose 131I treatments that could have been avoided by implementation of pre-therapy imaging based on result of post-therapy scintigraphy | Baseline and post-therapy
  In order to dertermine wheter a treatment could be considered futile a comparison between de I124-PET en post-therapy scan will be made and when the results are consistent we determine how many futile treatments could have been avoided when the I124 will be implemented in the future.

SECONDARY OUTCOMES:
Synchronised QA/QC of 124I-PET in the Netherlands | Before start study
  In order to make the scans quantifiable and comparable 124I-PET scans in this multicenter study a phantom study will be performed. The mean and median measured activity (Bq) in the different vials in the phantom will be assessed and compared to the known activity in the vial. In this way we will be able to create a calibration curve for each scanner.
- Translational correlation of 124I-PET and FDG-PET with histopathology (where available) and treatment outcome, in an explorative setting. | At follow-up
  - The outcome of the treatment is defined as a positive or negative post-therapy scan. This scan and both 124I-PET and FDG-PET will be correlated with histopathological features. The expression of different markers will be quantified in the samples. These results will also be compared with the results of the different scan modalities. In this way we aim to determine which histopathological features can predict outcome of the scans.
- To investigate whether 124I-PET has the same diagnostic, dosimetric and prognostic yield during stimulation with rhTSH and hormone withdrawal combined with low-iodine diet. | Baseline and during therapy
  Because 124I-PET will be performed both after stimulation with rhTSH and after withdrawal from levothyroxine it is possible to determine any differences in outcome from the two scan preparation strategies. Both visual assessment as the quantifiable data will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel PM Stokkel, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (15):
- Netherlands (15):
  - Rijnstate Hospital, Arnhem, Gelderland
  - UMC St. Radboud Nijmegen, Nijmegen, Gelderland
  - Bernard Verbeeten Institute, Tilburg, Noord-Braband
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Medical Center Alkmaar, Alkmaar, North Holland
  - St. Lucas Andreas Hospital, Amsterdam, North Holland
  - VUmc Medical Center, Amsterdam, North Holland
  - Medical spectrum Twente, Enschede, Overijssel
  - Isala Clinics, Zwolle, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden, South Holland
  - Meander Medical Center, Amersfoort, Utrecht
  - St. Antonius hospital, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Derived] Kist JW, de Keizer B, Stokkel MP, Hoekstra OS, Vogel WV; THYROPET study group. Recurrent differentiated thyroid cancer: towards personalized treatment based on evaluation of tumor characteristics with PET (THYROPET Study): study protocol of a multicenter observational cohort study. BMC Cancer. 2014 Jun 5;14:405. doi: 10.1186/1471-2407-14-405. PMID 24906384